CLINICAL TRIAL: NCT04104373
Title: The Ontario Neurodegenerative Disease Research Initiative
Acronym: ONDRI
Status: Completed | Type: Observational
Sponsor: Ontario Neurodegeneration Disease Research Initiative (Other)
Responsible Party: Sponsor
Other Study IDs: ONDRI2013
Record Dates: First submitted 2016-03-21; First posted 2019-09-26 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease; Amyotrophic Lateral Sclerosis; Frontotemporal Dementia; Parkinson Disease; Stroke
MeSH Terms: conditions — Alzheimer Disease; Amyotrophic Lateral Sclerosis; Frontotemporal Dementia; Parkinson Disease; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for genomic analysis of Deoxyribonucleic Acid (DNA) for rare variant genes potentially predictive of dementias.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Observational Cohort

SUMMARY:
The Ontario Neurodegenerative Disease Research Initiative (ONDRI) is a province-wide collaboration studying dementia and how to improve the diagnosis and treatment of neurodegenerative diseases including:

* Alzheimer's disease (AD)
* Parkinson's disease (PD)
* amyotrophic lateral sclerosis (ALS or Lou Gehrig's disease)
* frontotemporal lobar degeneration (FTD)
* vascular cognitive impairment, resulting from stroke (VCI)

DETAILED DESCRIPTION:
The Ontario Neurodegenerative Disease Research Initiative (ONDRI) is a research program designed to investigate similarities and differences of dementia among five diseases that will improve the diagnosis and treatment of neurodegeneration. The focus is on diseases that are associated with dementia: Alzheimer's disease/mild cognitive impairment, Parkinson's disease, amyotrophic lateral sclerosis (ALS or Lou Gehrig's disease), frontotemporal lobar degeneration, and vascular cognitive impairment (resulting from stroke).

ONDRI is a province-wide collaboration between more than 50 of Ontario's world-class neurodegenerative disease researchers and clinicians, four patient advocacy groups, the industrial sector, and more than 20 clinical, academic and research centres carried out in partnership with the Ontario Brain Institute (OBI).

Instead of only studying what's unique, our long-term observational study is seeking out the common early indicators and risk factors of the five diseases.

Our mandate is to ensure that the findings from the data collected are transformed into new diagnostic methods that will help detect diseases earlier, improved clinical practice that puts patients first, and eventually new effective treatments that will slow the diseases from progressing or even prevent the disease so people can continue to enjoy the later years of their lives.

More than 600 participants will be followed for up to three years and will complete assessments for genomics, gait and balance, eye measurements, neuropsychology, and neuroimaging and will donate their data to a comprehensive integrated data management system called Brain-CODE.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented.
* Participant must rate his/her level of proficiency in speaking and understanding English at 7 out of 10 or higher on the two LEAP-Q questions.
* Participant must have ≥ 8 years education.
* Participant with a minimum MoCA score of ≥18.

  * Exception: FTD minimum MoCA score of ≥ 14.
* Participant must have a reliable Study Partner. The Study Partner must:

  * Interact regularly with the participant (i.e., have contact with the participant at least once a month over the phone, email, or face-to-face);
  * Know the participant well enough to answer questions about the her/his cognitive abilities, communication skills, mood, and daily functioning (i.e., known the participant for at least 2 years);
  * Provide written informed consent and complete study questionnaires;
  * Be willing and able to assist in compliance with study procedures (if required).
* Geographic accessibility to the study site.
* Participant must be able to walk (assistive aids may be used, e.g., cane, walker, etc.).

Exclusion Criteria:

* Serious underlying disease other than the disease being studied which in the opinion of the investigator may interfere with the participant's ability to participate fully in the study.
* Any disease that would/could lead to death over the next 3 to 5 years (i.e., cardiac/renal/liver cancer) with poor prognosis.
* Participant has been diagnosed with more than one of the five diseases (AD/MCI, ALS, FTD, PD or VCI) being studied.
* History of alcohol or drug abuse, which in the opinion of the investigator, may interfere with the participant's ability to comply with the study procedures.
* Presence of any of the following clinical conditions:

  * Substance abuse within the past year.
  * Unstable cardiac, pulmonary, renal, hepatic, endocrine, hematologic, or active malignancy or infectious disease.
  * AIDS or AIDS-related complex.
  * Unstable psychiatric illness defined as psychosis (hallucinations or delusions) or untreated major depression within 90 days of the screening visit.
* Participant is currently enrolled in a disease modifying therapeutic (drug or interventional) trial or observational study that the Executive Committee feels would compromise study results.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately six hundred (600) participants who have one of the following diseases: VCI (150), AD/MCI (150); PD (150); FTD (60) and ALS (90) are to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Eye Tracking - Pro Saccade and Anti Saccade | 5 Years
  Pro-saccade task assesses simple sensory-motor function by following eye movement for specific tasks.
  • Anti-saccade task is identical to the pro-saccade task, except the instruction, indicated by fixation point (FP) colour,and is a sensitive indicator of cognitive disturbances.
Retinal Nerve Imaging | 5 years
  Institutions with the Heidelberg Spectralis with Ocular Coherence Tomography (OCT) Blue Peak Instrumentation will participate in this assessment.
  Both eyes of all participants will undergo:
  * Assessment of best corrected visual acuity
  * Digital colour fundus photography.
  * Retinal nerve imaging
Gait and Balance | 5 years
  All participants will perform walks along a 6 metre path while wearing hip and ankle accelerometers. Participants will perform three main tasks: 1) preferred walking speed, 2) dual task walking and 3) fast walking.
Genomics | 5 years
  Blood samples will be drawn by LifeLabs Medical Laboratory Services located in London, Ottawa, Toronto, Kingston, Thunder Bay, and Hamilton. Under extenuating circumstances, an appointment may be made with LifeLabs to have the blood samples drawn at home or in a residential facility.Samples must be drawn from Monday to Wednesday to allow for weekday shipping and receipt of samples at the OBI Biobank Sample Reception at Robarts Research Institute in London, Ontario (ON). LifeLabs standardized protocols for collection and overnight shipping will be followed. Subsequently, DNA aliquots for NeuroX microarray will be sent to Dr. Ekaterina Rogaeva at the University of Toronto in Toronto, ON. DNA aliquots for the OBI Neurodegeneration Re-sequencing Panel will remain with Dr. Robert Hegele at Robarts Research Institute in London, ON.
Neuropsychology | 5 years
  A battery of broad-based, standardized and validated cognitive assessments covering attention,memory, speech production, language and visuospatial function with a focus on coginitve domains reflection frontal network functioning and social attention. will be completed on an annual basis.
Neuroimaging | 5 years
  Imaging will be done on an annual basis to characterize the neuro-anatomical, microstructural, and functional profiles of dementia types and monitor changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Swartz, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (12):
- Canada (12):
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Providence Care Mental Health Services, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Parkwood Institute, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Elisabeth Bruyere, Ottawa, Ontario
  - Thunder Bay Regional Research Institute, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Baycrest, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected for the purpose of publications are to be shared via a controlled public release along with the accompanying data dictionaries and other supplementary files. All data shared are de-identified in accordance with the policies set out by the Ontario Brain Institute (OBI).
Time Frame: Initial data release of Baseline data was made available June 8, 2022. Further release of longitudinal data and raw, de-identified neuroimaging data will be made available on September 30, 2023.
Access Criteria: Access to data is provided to users with an affiliation with an accredited academic institution, think tank, company, or other research organization. Users must also submit a Data Access Request along with Research Ethics Board approval which are then reviewed and approved by OBI's data access committee.
URL: https://indocconsortium.atlassian.net/wiki/spaces/JSDNXT/pages/1933279255/Data+Release+Articles

REFERENCES:
- [Derived] Ryoo SW, Lin WZ, Magliocco A, Ruthirakuhan M, Wong YY, Perfetto SE, Huang C, Anita NZ, Arnott SR, Lang AE, Symons S, Hegele RA, Goubran M, Ramirez J, Ottoy J, Rabin JS, MacIntosh BJ, Lanctot KL, Liang N, Cogo-Moreira H, Taha AY, Swardfager W; ONDRI Investigators. Metabolic and vascular contributions to dementia: Soluble epoxide hydrolase-derived linoleic acid oxylipins and glycemic status are related to cerebral small vessel disease markers, atrophy, and cognitive performance. Alzheimers Dement. 2025 Oct;21(10):e70718. doi: 10.1002/alz.70718. PMID 41059602